CLINICAL TRIAL: NCT00479245
Title: WHODAS-II for Patients With Nonspecific Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate, lower than expected. Organizational changes made it impossible for recruiting centers to continue
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FK-R-17
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; disability; fear avoidance beliefs; quality of life
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule)
  Interventions: Other: Set of questionnaires (respondent)

INTERVENTIONS:
Other: Set of questionnaires (respondent) — To determine the measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule)

SUMMARY:
The main purpose of this study is to determine the measurement characteristics of WHODAS-II (World Health Organization Disability Assessment Schedule), as well as to analyze its correlation with low back pain (Visual Analog Scale, VAS), disability (Spanish version of the Roland Morris Questionnaire, RMQ), fear avoidance beliefs and attitudes (Spanish version of the FAB Questionnaire, FABQ) and quality of life (SF-12). Measurements will be taken at baseline and 6 days later (day 7).

ELIGIBILITY:
Inclusion Criteria:

* Patients seen for nonspecific low back pain, with or without referred pain
* Able to read and write
* Have signed the informed consent form

Exclusion Criteria:

* Central nervous system pathology (with or without treatment)
* Diagnosis of rheumatic inflammatory disease or fibromyalgia
* Red flags for underlying systemic disease
* Criteria for diagnosis of symptomatic herniated disc or symptomatic spinal stenosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement characteristics of WHODAS-II | At baseline and at 7 days

SECONDARY OUTCOMES:
Correlation between WHODAS-II and VAS, RMQ, FABQ and SF-12 in nonspecific low back pain | At baseline and at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; José Luis Peña, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

REFERENCES:
- [Background] Bombardier C. Outcome assessments in the evaluation of treatment of spinal disorders. Introduction. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3097-9. doi: 10.1097/00007632-200012150-00002. No abstract available. PMID 11124723
- [Background] Chwastiak LA, Von Korff M. Disability in depression and back pain: evaluation of the World Health Organization Disability Assessment Schedule (WHO DAS II) in a primary care setting. J Clin Epidemiol. 2003 Jun;56(6):507-14. doi: 10.1016/s0895-4356(03)00051-9. PMID 12873644
- [Background] van Tubergen A, Landewe R, Heuft-Dorenbosch L, Spoorenberg A, van der Heijde D, van der Tempel H, van der Linden S. Assessment of disability with the World Health Organisation Disability Assessment Schedule II in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Feb;62(2):140-5. doi: 10.1136/ard.62.2.140. PMID 12525383